CLINICAL TRIAL: NCT04507451
Title: Inspiratory and Expiratory Muscle Training in Critically Ill Patients Weaned From Mechanical Ventilation
Brief Title: Respiratory Muscle Training in ICU Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Rousseau, Head of clinic, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RESP-USI
Record Dates: First submitted 2020-08-01; First posted 2020-08-11 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Critical Illness; Inspiratory Muscle Strength; Mechanical Ventilation; Respiratory Muscle Training
MeSH Terms: conditions — Critical Illness | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant
Masking Description: patients are masked: they will all benefit from respiratory physiotherapy, with placebo or real muscle training investigator and care providers are unmasked, as they set the training parameters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trained group (Experimental): Patients will benefit from usual respiratory physiotherapy (secretion clearance treatment and recruitment maneuvers), and muscle training. This program will be delivered 5 days a week.
  Inspiratory muscle training (IMT): using a threshold IMT device with mouthpiece, 5 sets of 6 breaths, intensity is prescribed at 60% of maximal inspiratory pressure for the first set, and then increased to the highest tolerable intensity to allow completion of the 6th breath Expiratory muscle training (EMT): using a bottle filled with water, starting at 5cm and then increased to 8 cm gradually, 5 sets of 6 breaths
  Training program starts after mechanical ventilation weaning, as soon as the patient is collaborative, and is continued until 1 month after ICU discharge
  Interventions: Procedure: inspiratory and expiratory muscle training
- Untrained group (Placebo Comparator): Patients will benefit from usual respiratory physiotherapy (secretion clearance treatment and recruitment maneuvers), and muscle exercises that are not planned to train muscles. This program will be delivered 5 days a week.
  Inspiratory exercises: fractionated inspiration, 5 sets of 6 breaths Expiratory exercises: using a bottle filled with water (1 cm)
  Exercises program starts after mechanical ventilation weaning, as soon as the patient is collaborative, and is continued until 1 month after ICU discharge
  Interventions: Procedure: inspiratory and expiratory exercises

INTERVENTIONS:
Procedure: inspiratory and expiratory muscle training — inspiratory muscle training using threshold IMT device expiratory muscle training using a bottle filled of water
  Arms: Trained group
Procedure: inspiratory and expiratory exercises — inspiratory exercise using fractionated inspirations expiratory exercise using a bottle filled with water at a minimum level
  Arms: Untrained group

SUMMARY:
Respiratory muscle weakness is common after mechanical ventilation and occurs early. This can limit functional recovery. Respiratory muscle training is often neglected in clinical practice. Some data indicates that inspiratory muscle training increases inspiratory muscle strength and quality of life. The aim of the study is to assess the impact of combined inspiratory and expiratory muscle training on inspiratory muscle strength. The second aim is to assess the impact of this training program on expiratory muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* patient from mechanical ventilation after at least 24 hours of support
* collaborative patient

Exclusion Criteria:

* confusion, mental disorder
* not french speaking
* pulmonary surgery in the past 12 months
* external ventricular drain
* previous pneumothorax or pneumothorax not drained
* rib fractures
* alveolar hemorrhage
* hemodynamic instability
* labial occlusion impossible (face burn, facial paralysis)
* patient refusal

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
change in inspiratory muscle strength | between 7 to 15 days after ICU discharge (compared to ICU discharge)
  measurement of maximal inspiratory pressure
change in inspiratory muscle strength | 1 month after ICU discharge (compared to ICU discharge)
  measurement of maximal inspiratory pressure

SECONDARY OUTCOMES:
change in expiratory muscle strength | between 7 to 15 days after ICU discharge (compared to ICU discharge)
  measurement of maximal expiratory pressure
change in expiratory muscle strength | 1 month after ICU discharge (compared to ICU discharge)
  measurement of maximal expiratory pressure
respiratory infections | 1 month after ICU discharge
  number of respiratory infections requiring antibiotics after ICU discharge
change in dyspnea perception | 1 month after ICU discharge (compared to hospital discharge)
  assessed using Dyspnea-12 questionnaire (score from 0 to 36, 36 indicating a maximal dyspnea)
impact of dyspnea on physical activities | between 7 to 15 days after ICU discharge
  assessed using modified Medical Research Council (m-MRC) score: stage 0 to 4 (last stage indicating a patient too dyspneic to leave house or breathless when dressing)
impact of dyspnea on physical activities | 1 month after ICU discharge
  assessed using modified Medical Research Council (m-MRC) score: stage 0 to 4 (last stage indicating a patient too dyspneic to leave house or breathless when dressing)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No